CLINICAL TRIAL: NCT03262987
Title: Color Doppler U/S vs MSCT Venography in the Diagnosis of May-Thurner Syndrome
Brief Title: Color Doppler U/S vs MSCT Venography in May-Thurner Syndrome
Acronym: USvsCTV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Gamal Mokhtar, Resident Doctor, Assiut University
Other Study IDs: May-Thurner Syndrome
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: May-Thurner Syndrome
MeSH Terms: conditions — May-Thurner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
May-Thurner syndrome is the result of compression of the left common iliac vein between the right common iliac artery and overlying vertebrae.

In This Study , We will detect the role of color doppler US in the diagnosis of May-Thurner Syndrome in comparison to Direct CT Venography

DETAILED DESCRIPTION:
May-Thurner syndrome (MTS) is a venous compression syndrome in which the left common iliac vein is compressed between the lower lumbar spine and the right common iliac artery. While asymptomatic compression is very common, the process can lead to morbidity in selected individuals, most commonly deep venous thrombosis (DVT) and the sequelae thereof. Radiologists must recognize the diagnosis because of the unique management, which differs from DVT without iliac vein compression.

The most common clinical presentation is unilateral leg swelling due to acute DVT. It can also present as chronic venous insufficiency or chronic thrombosis with symptoms of venous hypertension and venous stasis namely claudication, pain, swelling, varicose veins and / or ulceration.

Conventional invasive catheter venography remains the gold standard for diagnosis,but the decision to undertake invasive venography should be made only after reviewing all available clinical data and alternative, less invasive imaging options have been exhausted.

When visualization of the common iliac veins is possible, MTS may be diagnosed with transabdominal color Doppler U/S.

MDCT with IV contrast is a fast, widely available examination for the diagnosis of MTS and accompanying complications .

Magnetic resonance imaging (MRI) with MR venography is an attractive modality for the diagnosis, However, MRI is expensive, time consuming, has more limited availability than computed tomography (CT) and ultrasound, and may be impossible in select patients.

ELIGIBILITY:
Inclusion Criteria:

* advanced chronic venous insufficiency submitted to clinical treatment for at least 1 year with no response.
* Subject must be > 18 and < 80 years of age.
* informed consent document before the planned procedure.
* On duplex ultrasound: patent common femoral vein, and patent deep femoral vein, and/or femoral vein of the study leg.

Exclusion Criteria:

* Previous venous stent implantation involving the study leg or inferior vena cava
* Previous venovenous bypass surgery involving the study leg
* Known reaction or sensitivity to iodinated contrast that cannot be managed with premedication.
* Subjects who are pregnant (women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment).
* Acute deep venous thrombosis involving either leg.
* Known history of chronic total occlusion of the common femoral vein of the study leg.
* Venous compression caused by tumor encasement.
* Venous outflow obstruction caused by tumor thrombus.
* Elevated baseline blood creatinine (value greater than the upper limit of the normal range).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients suffering from advanced chronic venous insufficiency in the left leg.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Color Doppler U/S Vs MSCT Venography in the diagnosis of May-Thurner Syndrome | 1 year
  Determine the sensitivity, specificity and accuracy of non invasive color doppler ultrasound, using direct and indirect ultrasonographic signs, in the diagnosis of May-Thurner Syndrome , considering direct CT Venography as the gold standard for this diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Koraim, Ass. Prof., Study Chair — Assiut university, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
to be shared when finished